CLINICAL TRIAL: NCT04059276
Title: Functional, Structural, and Metabolic Central Nervous System Changes Following Damage of the Central Nervous System
Brief Title: CNS Changes Following Stroke
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00937 - Stroke
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with stroke
  Interventions: Diagnostic Test: MRI
- Healthy subjects
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — We will examine chronic (>3 months post stroke) patients using functional, structural, and metabolic MRI in both the brain and the spinal cord.
  Groups: Patients with stroke
Diagnostic Test: MRI — We will examine healthy control participants using functional, structural, and metabolic MRI in both the brain and the spinal cord.
  Groups: Healthy subjects

SUMMARY:
The objective of this study is to better understand the structural and functional changes that the CNS undergoes following stroke and how these changes relate to clinical measures. Both macroscopic and microscopic changes of the brain and the spinal cord will be examined in stroke patients and compared to healthy controls. In terms of structural plasticity, we aim to identify MR biomarkers that allow predicting the course of the patient's neurological status and accurately describe the course of the disease and the recovery. Importantly, we aim to investigate which factors scale the patients' symptoms.

In terms of functional plasticity, we will combine fMRI with behavioural motor and sensory testing to understand i) the structural and functional interplay between spinal and supraspinal neural circuits after stroke possibly driven by beneficial plasticity/regeneration vs. maladaptive plasticity/degeneration and ii) which clinical and behavioural determinants drive functional hand representations in the primary somatosensory and motor cortices to be maintained and which determinants drive reorganisation of functional representations following sensory input loss. We will further investigate the contribution of brainstem reorganisation to plasticity observed at the cortical level and, by doing so, aim to better understand the mechanistic underpinnings of functional reorganisation.

ELIGIBILITY:
Inclusion Criteria - Patients:

* Age 18-80
* Stroke (> 3months)
* Signed informed consent

Exclusion Criteria - Patients:

* Contraindications to magnetic resonance imaging
* Neurological impairment of body function impairments not induced by stroke
* BMI > 40
* Pregnancy
* Claustrophobia

Inclusion Criteria - Healthy subjects:

* Age 18-80
* Signed informed consent

Exclusion Criteria - Healthy subjects:

* Contraindications to magnetic resonance imaging
* Pregnancy
* Neurological illness
* Impairment of body function induced by stroke
* Claustrophobia
* BMI >40

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with stroke and healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Conventional magnetic resonance imaging (MRI) parameter | Up to 50 weeks]
  Structural characteristics in the brain and spinal cord are assessed in chronic stroke patients using conventional MRI and compared to healthy controls

SECONDARY OUTCOMES:
Magnetic resonance spectroscopy (MRS) parameter | Up to 50 weeks
  Metabolic parameter are assessed in chronic stroke patients using MRS in the brain and spinal cord and compared to healthy controls
Functional MRI (fMRI) parameter | Up to 50 weeks
  Brain activity or change of brain activities between 2 to 5 time points is assessed using fMRI during resting-state or a specific task in chronic stroke patients and compared to healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Freund, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland